CLINICAL TRIAL: NCT02043119
Title: BEST ABCs: Benefits and Effectiveness of Support Offered Through A Breastfeeding Clinic Study
Acronym: BEST ABCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20130560-01H; 13/31E (Other: CHEO REB)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Exclusive Breastfeeding Rates; Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breastfeeding Clinic (Active Comparator): A breastfeeding clinic that mothers can attend with their infants up to one month post delivery.
  Interventions: Behavioral: Breastfeeding Clinic
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Breastfeeding Clinic
  Arms: Breastfeeding Clinic

SUMMARY:
Currently, healthy mothers willing to breastfeed their babies are discharged from the hospital on an average 2 days after a vaginal delivery or 3.5 days after a C-section, at a time where breastfeeding is far to be well established. Following discharge, women can access breastfeeding support from Public Health Units, lactation consultants, health care providers, and Internet (e.g. from breastfeeding associations). Despite the current support, duration and exclusivity rates of breastfeeding drop precipitously in the first weeks and months after birth.

We have obtained funding from the Ontario Ministry of Health and Long Term Care to evaluate the efficacy and cost effectiveness of a post-partum clinic based in the community. This clinic, staffed by a family physician (in the morning), a registered nurse and a lactation consultant, will provide breastfeeding support during the first month after delivery as well as ensure a safe transition from hospital to the community for mothers and newborn babies. The clinic, affiliated with TOH, will be found at Harmony Medical Centre, 152 Cleopatra Drive, located south-west of downtown, a 15 minute drive from the Civic campus and 20 minutes from the General campus. The Harmony Clinic has abundant parking (free on the street or a small fee inside the associated lot) and is fully accessible.

In its initial phase, the future clinic would enroll only women willing to participate in a research program to evaluate this new program. The clinic will be opening in November 2013 and currently (July - October 2013) we are conducting a pilot study to test feasibility of recruitment and test the surveys and database for this project. Women will be recruited at the Ottawa Hospital (General and Civic campus) and randomized to either receive standard-care or to be given access to the post-partum clinic and be discharged within approximately 24 hours following a vaginal delivery or 48 hours following a C-section. They will have an appointment booked at the breastfeeding clinic within 48 hours after discharge for maternal and neonatal care as well as breastfeeding support. Enrolled women will have access to additional clinic visits for one month after delivery. Information will be collected from their medical chart as well as through surveys that will be sent to them at 15 days, 30 days and 3 months after delivery. We will compare the data and information on the experience of women who attended the breastfeeding clinic and those who did not attend the clinic. With this data we will be able to determine if this type of breastfeeding clinic is beneficial to new mothers and their newborn babies and if it really does increase the exclusive breastfeeding rate at 3 months (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Mothers having delivered a baby at The Ottawa Hospital - General or Civic Campus:

  1. Who are ≥ 18 years at the time of enrollment
  2. Who are any parity, with a singleton infant born > 36 + 6 weeks of Gestational Age
  3. Who have no medical counter indication for discharge at 24 (±12) hours post vaginal delivery or 48 (±12) hours post C-section delivery and for which the physician (family physician or obstetrician) has agreed that the mother is eligible
  4. Who are breastfeeding and intend to breastfeed their baby upon discharge
  5. Whose infant is healthy with no counter indication for discharge at 24 (±12) hours post vaginal birth or 48 (±12) hours post C-section birth and for which the physician (family physician or paediatrician) has agreed that the infant is eligible
  6. Who can be contacted by phone or E-mail after hospital discharge

Exclusion Criteria:

* Mothers:

  1. Who have had breast surgery
  2. Who do not understand French or English
  3. Who are unable to present to the clinic (transport not available)
  4. Who have birthed multiples or preterm
  5. Whose infants are exclusively formula-fed
  6. Who are adoptive mothers
  7. Who have been identified with a psychological risk that may impede her ability to attend the first appointment at the clinic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The rate of exclusive breastfeeding at 3 months post-birth. | 3 months post birth
  The rate of exclusive breastfeeding at 3 months post-birth. We define exclusive breastfeeding as the feeding of the infant's mother's milk only for at least 2 weeks prior to collected outcome.

SECONDARY OUTCOMES:
Rates of hyperbilirubinemia requiring phototherapy or hospitalization | 6 months
Poor infant weight gain requiring intervention (pumping, supplementation, hospitalization) | 24 hours - 3 months
Incidence of breastfeeding difficulties (e.g., sore nipples, insufficient milk supply, inadequate latch, engorgement) | 24 hours - 3 months
Breastfeeding self efficacy score (Breastfeeding Self Efficacy Scale or BSES) at 2 weeks, 1 month and 3 months | 2 weeks, 1 month, 3 months
Score of the Edinburgh Post-partum Depression Scale for new mothers | 3 weeks
Access to community-based services: Public Health Clinics, Family Doctor, Pediatrician | 2 weeks, 1 month, 3 months
Number of emergency department visits for the mother and the baby | 6 months
Number of hospital readmissions for the mother and her baby | 6 months
Mothers' satisfaction with the support received | 3 months
Length of stay in the hospital, from delivery to discharge | 2 weeks
Costs associated with this community-based postpartum clinic | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lacaze-Masmonteil, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Gavine A, Shinwell SC, Buchanan P, Farre A, Wade A, Lynn F, Marshall J, Cumming SE, Dare S, McFadden A. Support for healthy breastfeeding mothers with healthy term babies. Cochrane Database Syst Rev. 2022 Oct 25;10(10):CD001141. doi: 10.1002/14651858.CD001141.pub6. PMID 36282618
- [Derived] Laliberte C, Dunn S, Pound C, Sourial N, Yasseen AS 3rd, Millar D, Rennicks White R, Walker M, Lacaze-Masmonteil T. A Randomized Controlled Trial of Innovative Postpartum Care Model for Mother-Baby Dyads. PLoS One. 2016 Feb 12;11(2):e0148520. doi: 10.1371/journal.pone.0148520. eCollection 2016. PMID 26871448